CLINICAL TRIAL: NCT05549219
Title: A Phase 2, Randomized, Open-Label, 24-Week Study to Assess the Pharmacodynamics, Safety, Tolerability, and Pharmacokinetics of Multiple Doses of GLM101 Administered Intravenously to Adult, Adolescent, and Pediatric Participants With PMM2-CDG
Brief Title: 24-Week Study to Assess the PD, Safety, Tolerability, and PK of GLM101 in Participants With PMM2-CDG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glycomine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GLM101-002
Record Dates: First submitted 2022-08-24; First posted 2022-09-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pmm2-CDG; Phosphomannomutase 2 Deficiency
Keywords: Pmm2-CDG; Pmm2; CDG; GLM101
MeSH Terms: conditions — Congenital disorder of glycosylation type 1A

STUDY DESIGN:
Intervention Model Description: Participants will randomized to receive either 10 mg/kg GLM101 or 20 mg/kg GLM101. Subsequently, if safety and tolerability are demonstrated at 10 and 20 mg/kg, 30 mg/kg groups will be added.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 10 mg/kg GLM101 (Experimental): GLM101 IV infusions, given weekly
  Interventions: Drug: GLM101
- 20 mg/kg GLM101 (Experimental): GLM101 IV infusions, given weekly
  Interventions: Drug: GLM101
- 30 mg/kg GLM101 (Experimental): GLM101 IV infusions, given weekly
  Interventions: Drug: GLM101

INTERVENTIONS:
Drug: GLM101 — GLM101 IV Infusion

SUMMARY:
This is a Phase 2, randomized, open-label, 24-week treatment study to evaluate the potential pharmacodynamic (PD) activity, safety, tolerability, and pharmacokinetics (PK) of GLM101 in adult, adolescent, and pediatric, patients with a confirmed diagnosis of PMM2-CDG. The planned doses of GLM101 to be investigated are 10, 20, and 30 mg/kg. The study will consist of a Screening Period, a 24-week (6-month) Treatment Period, and a 30-day (1-month) Follow-Up Period.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female, 18 to 65 years of age, inclusive, at Screening (Cohorts 1-3, 7), 12-17 years of age, inclusive, at Screening (Cohort 4) or 2-11 years of age, inclusive, at Screening (Cohorts 5 and 6);
* Molecularly confirmed diagnosis of PMM2-CDG. Diagnosis is defined as biallelic pathogenic and/or likely pathogenic variants, or, in the case of variants of uncertain pathogenicity, demonstration of bi-allelic variants AND phosphomannomutase-2 (PMM2) enzyme activity consistent with a diagnosis of PMM2-CDG. Historical diagnosis with lab report(s) on file is permitted;
* If the participant is a female of childbearing potential (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile (permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy)) she must not be pregnant (confirmed by a negative serum pregnancy test), is using a medically accepted method of contraception (abstinence, a hormonal contraceptive associated with inhibition of ovulation in conjunction with a barrier method, or use of an intrauterine device), and must agree to continue using this method for 50 days after the last infusion of GLM101; Note: sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception;
* If the participant is a female of non-childbearing potential, she must be pre-pubertal, surgically sterile, or must have an ovarian dysfunction confirmed by a follicle stimulating hormone (FSH) >40 IU/L and absence of menses for 12 months without an alternative medical cause;
* If the participant is a sexually active male with female partners, the sexually mature, nonsterile male participant agrees to use a medically acceptable method of contraception (abstinence, the partner taking a hormonal contraceptive in conjunction with a male condom, or use by the partner of an intrauterine device with a male condom) and agrees to continue using this method for 50 days after the last infusion of GLM101. Males are considered surgically sterile if they have undergone bilateral orchiectomy or vasectomy at least 3 months prior to Screening;
* If the participant is male, he must agree to refrain from donating sperm during the study and 50 days after the last infusion of GLM101;
* Is willing and able to provide informed consent/assent, directly or through his/her legally authorized representative.

Exclusion Criteria:

* Diagnosis of congenital disorder of glycosylation (CDG) other than PMM2; Diagnosis is defined as biallelic pathogenic and/or likely pathogenic variants, or, in the case of variants of uncertain pathogenicity, demonstration of bi-allelic variants AND the defined CDG enzyme activity consistent with a diagnosis of the CDG other than PMM2 CDG.
* Has an active infection requiring parenteral antibiotics, antivirals, or antifungals or treatment with systemic steroids within 7 days prior to Screening;
* Has confirmed active coronavirus disease-2019 (COVID-19) or tests positive for severe acute respiratory syndrome coronavirus 2 (SARS CoV 2) at Screening or check in to the clinical site;
* ALT or AST >3× ULN OR total bilirubin >2× ULN or INR >1.5
* Has a history of a severe allergic reaction to any drug or excipients of GLM101 (as listed in the GLM101 Investigator's Brochure);
* Has a known history of poor venous access;
* Has a history of liver transplant;
* Has a history of drug or alcohol use disorder within 12 months prior to Screening;
* Has had a major surgical procedure within 30 days prior to Screening;
* Has Screening or eligibility confirmation laboratory value(s) outside the laboratory reference range considered clinically significant and not related to PMM2-CDG;
* If female, has a positive serum pregnancy test during Screening;
* If female, must not be breastfeeding;
* Has serology positive for hepatitis B surface antigen or hepatitis C antibody during Screening;
* Has history or presence, upon clinical evaluation, of any illness that might impact the safety of GLM101 infusion or evaluability of drug effect based on the Investigator's and Medical Monitor's discretion;
* Has a QTc ≥ 450 ms, or other clinically significant ECG abnormalities;
* Has uncontrolled cardiovascular, hepatic, pulmonary, gastro-intestinal, endocrine, metabolic, ophthalmologic, immunologic, psychiatric or other significant disease;
* Is currently participating in another interventional clinical study or has completed another clinical study with an investigational drug or device within 30 days or 5 half-lives before GLM101 infusion.
* Weight exceeds 75 kg.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Evaluate changes from baseline in ataxia | 12 weeks and 24 weeks
  Changes in ICARS (International Co-operative Ataxia Rating Scale)

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events assessed by severity and frequency | 12 weeks and 24 weeks
  Evaluate Safety and tolerability of multiple doses of GLM101. Collection and assessment of adverse events, adverse event of special interest, serious adverse events, deaths, discontinuations, clinical laboratory tests, vital signs and physical exam.
Maximum observed plasma concentration (Cmax) | over 24 weeks
  Assessment of the pharmacokinetics (PK) of GLM101
Time to maximum observed plasma concentration (Tmax) | over 24 weeks
  Assessment pharmacokinetics (PK) of GLM101
Area under the plasma concentration vs. time curve (AUC) | over 24 weeks
  Assessment of the pharmacokinetics (PK) of GLM101

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Clinical Research of West Florida, Tampa, Florida
  - Mayo Clinic, Rochester, Minnesota
- Hospital Sant Joan de Déu, Barcelona, Spain
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No